CLINICAL TRIAL: NCT03448822
Title: Sentinel Lymph Node Procedure in Testicular Germ Cell Tumour
Acronym: SENATOR
Status: Not yet recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: M18TGC
Record Dates: First submitted 2018-01-30; First posted 2018-02-28 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-01

CONDITIONS: Testicular Germ Cell Tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sentinel node procedure: a robot-assisted laparoscopic sentinel node procedure.
  Interventions: Procedure: sentinel node procedure

INTERVENTIONS:
Procedure: sentinel node procedure — a robot-assisted laparoscopic sentinel node procedure to detect occult lymph node metastasis

SUMMARY:
Assessment of accuracy of sentinel node biopsy, defined as the false negative rate.

DETAILED DESCRIPTION:
Current practice in patients with Clinical Stage I (CS I) testicular germ cell tumour is active surveillance after orchiectomy, with relapses occurring in 15-20% of patients. The majority of relapses occur in the lymph nodes as lymphogenic spread is the dominant route of dissemination. A sentinel node procedure, in which the sentinel lymph node is resected and pathologically examined, could be more reliable to identify patients who are likely to relapse.

Early identification of patients with micro-metastases in the sentinel node makes it possible to treat these patients at the earliest possible moment. Absence of metastases could lead in the future to a less intensive follow up protocol than the present one.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of testicular germ cell tumour, based on physical examination, ultrasound imaging, and tumour markers
* Patients 18 years and older
* No evidence of metastases on first staging (thoraco-abdominopelvic CT)
* Written and signed informed consent

Exclusion Criteria:

* Patients with evidence of metastases at first staging
* Patients with a second primary tumour
* Patients with recent (< 6 months before diagnosis) surgical treatment to the external genitals or recent surgical intervention in the inguinal or retroperitoneal regions
* Patients with previous abdominal surgery, necessitating open surgical approach for the sentinel node biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — testical germ cell tumors
Study Population: Patients suspected of testicular germ cell tumour
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
identify patients witha low risk of cancer recurrenceincluded in current active surveillance protocols. | surgery 1 day, follow up 5 years
  identify patients who have such a low risk of cancer recurrence that it is not necessary anymore to be included in current active surveillance protocols by removing the sentinal lymph node to check for occult metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Simon Horenblas, MD, PhD, Principal Investigator — NKI-AvL